CLINICAL TRIAL: NCT02457377
Title: Laparoscopic Transabdominal Cerclage: A New Ideal Approach
Brief Title: Laparoscopic Transabdominal Cerclage: New Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Maged (Other)
Responsible Party: Sponsor-Investigator, Ahmed Maged, Assistant professor, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 136
Record Dates: First submitted 2015-05-25; First posted 2015-05-29 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Recurrent Abortion
Keywords: recurrent abortion; cerclage; laparoscopy; cervical imcompetence
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic cerclage (Experimental): The vesico-uterine peritoneum is opened & the urinary bladder is dissected downwards . Both needles are passed through the lower uterine tissue medial to uterine vessels on the right & left sides . Then, both needles are passed through the remaining cervical tissue medial to uterosacral ligaments towards the posterior vaginal fornix (on the right & left sides) guided by laparoscopic illumination . When the needles' blunt ends pierce the vaginal vault, the assistant pull them through the posterior vaginal fornix . After trimming of both needles, the Mersilene tape is tied tightly behind the intravaginal segment of the cervix with five knots &
  Interventions: Procedure: laparoscopic cerclage

INTERVENTIONS:
Procedure: laparoscopic cerclage — The vesico-uterine peritoneum is opened & the urinary bladder is dissected downwards . Both needles are passed through the lower uterine tissue medial to uterine vessels on the right & left sides . Then, both needles are passed through the remaining cervical tissue medial to uterosacral ligaments towards the posterior vaginal fornix (on the right & left sides) guided by laparoscopic illumination . When the needles' blunt ends pierce the vaginal vault, the assistant pull them through the posterior vaginal fornix . After trimming of both needles, the Mersilene tape is tied tightly behind the intravaginal segment of the cervix with five knots &

SUMMARY:
A 5-mm non-absorbable Mersilene polyester suture, with adjacent partially straightened blunt needles, is introduced into the abdominal cavity through the 5-mm trocar. However, flattening the curvature of the needles, while introducing the tape into the abdomen, will eventually pose a challenge during placement of the stitch (the needles' curvatures guarantee that the tissue penetration is done away from the uterine vessels).

To overcome this problem, the following method was devised. A one cm suprapubic incision is made on the abdomen with a scalpel short of the peritoneum. A needle holder loaded with the needle is pushed through the incision until the tip is seen inside the peritoneal cavity. A grasper from one of the flank ports receives the tip and the needle is delivered carefully (FIGURE 1). The rest of the tape is pulled until the blunt end of the other needle appears, to be delivered in the same way but in the reverse order.

• Operative Steps The vesico-uterine peritoneum is opened using scissors & the urinary bladder is dissected downwards from the lower uterine segment to expose the uterine vessels anteriorly on both sides . Both needles are passed through the lower uterine tissue medial to uterine vessels on the right & left sides (from anterior to posterior) . Then, both needles are passed through the remaining cervical tissue medial to uterosacral ligaments towards the posterior vaginal fornix (on the right & left sides) guided by laparoscopic illumination . When the needles' blunt ends pierce the vaginal vault, the assistant pull them through the posterior vaginal fornix . After trimming of both needles, the Mersilene tape is tied tightly behind the intravaginal segment of the cervix with five knots & the ends of the stitch are trimmed. The vesico-uterine peritoneum is then reapproximated over the laparoscopic cerclage with a running (00) Monocryl suture that is tied intracorporeally.

DETAILED DESCRIPTION:
Under general anaesthesia, the patient is placed in the modified dorsal lithotomy position. The patient is then prepped and draped in the usual fashion for an abdominal & vaginal procedure. A vaginal speculum is inserted into the vagina to expose both the cervix and posterior fornix. A uterine manipulator is inserted in the uterus in non-pregnant patients, followed by placement of a Foley's catheter in the bladder. As regards port placement, a 10-mm umbilical trocar & two 5-mm trocars in right & left lower quadrants are inserted.

• Introduction of Mersilene Tape into the Abdominal Cavity: A 5-mm non-absorbable Mersilene polyester suture, with adjacent partially straightened blunt needles, is introduced into the abdominal cavity through the 5-mm trocar. However, flattening the curvature of the needles, while introducing the tape into the abdomen, will eventually pose a challenge during placement of the stitch (the needles' curvatures guarantee that the tissue penetration is done away from the uterine vessels).

To overcome this problem, the following method was devised. A one cm suprapubic incision is made on the abdomen with a scalpel short of the peritoneum. A needle holder loaded with the needle is pushed through the incision until the tip is seen inside the peritoneal cavity. A grasper from one of the flank ports receives the tip and the needle is delivered carefully . The rest of the tape is pulled until the blunt end of the other needle appears, to be delivered in the same way but in the reverse order.

• Operative Steps The vesico-uterine peritoneum is opened using scissors & the urinary bladder is dissected downwards from the lower uterine segment to expose the uterine vessels anteriorly on both sides . Both needles are passed through the lower uterine tissue medial to uterine vessels on the right & left sides (from anterior to posterior) Then, both needles are passed through the remaining cervical tissue medial to uterosacral ligaments towards the posterior vaginal fornix (on the right & left sides) guided by laparoscopic illumination . When the needles' blunt ends pierce the vaginal vault, the assistant pull them through the posterior vaginal fornix . After trimming of both needles, the Mersilene tape is tied tightly behind the intravaginal segment of the cervix with five knots & the ends of the stitch are trimmed. The vesico-uterine peritoneum is then reapproximated over the laparoscopic cerclage with a running (00) Monocryl suture that is tied intracorporeally.

ELIGIBILITY:
Inclusion Criteria:

* Failed vaginal cerclage 2 successive spontaneous mid trimesteric abortion

Exclusion Criteria:

* rupture of membranes Uterine contractions evidence of intraamniotic infections contraindications to laparoscopy

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2004-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
completing pregnancy | 36 weeks of gestation
  number of participants with completing pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt